CLINICAL TRIAL: NCT03805945
Title: Effects of Dexmedetomidine on Mood and Breastfeeding in Parturient Undergoing Elective Cesarean Section.
Brief Title: Effect of Dexmedetomidine on Parturient Undergoing Elective Cesarean Section.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XYFY2019-KL054-02
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-01

CONDITIONS: Cesarean Section
Keywords: Cesarean Section; Dexmedetomidine; Breast Feeding; Recovery quality
MeSH Terms: conditions — Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine group (Experimental): After umbilical cord was cut, a loading dose of dexmedetomidine was pumped at 0.5ug/kg within 10min, followed by a further infusion of dexmedetomidine at 0.5ug /kg/h until the end of the surgery.Then connected with patient-controlled intravenous analgesia pump (dexmedetomidine 2ug/kg + sufentanil 1.5ug/kg + dolasetron 25mg/100ml saline).
  Interventions: Drug: dexmedetomidine group
- control group (Placebo Comparator): Continuous infusion of saline after the umbilical cord was cut until the end of the operation.Then connected with patient-controlled intravenous analgesia pump (sufentanil 1.5ug/kg + dolasetron 25mg/100ml saline).
  Interventions: Drug: control group

INTERVENTIONS:
Drug: dexmedetomidine group — After the fetus was delivered, low-dose dexmedetomidine intraoperative infusion, postoperative low-dose dexmedetomidine patient-controlled intravenous analgesia pump(the background infusion is 2 ml/h, the bolus dose is 0.5 ml, the lock time is 15 min).
  Other Names: D group
  Arms: dexmedetomidine group
Drug: control group — After the fetus was delivered, saline intraoperative infusion, postoperative patient-controlled intravenous analgesia pump(the background infusion is 2 ml/h, the bolus dose is 0.5 ml, the lock time is 15 min) without dexmedetomidine.
  Other Names: C group
  Arms: control group

SUMMARY:
The purpose of this study was to investigate whether dexmedetomidine used in the perioperative period of elective cesarean section can improve maternal mood, improve analgesic effect, improve maternal recovery quality, and then make the breastfeeding better.At the same time, this experiment attempts to explore the optimal dose of dexmedetomidine to produce the above effect.

DETAILED DESCRIPTION:
After obtaining the informed consent, parturients were randomly divided into two groups according to the computer-generated random number table, namely, dexmedetomidine group and the control group.Spinal anesthesia is administered to all maternal women undergoing elective cesarean delivery. Immediately after the umbilicus is cut, the infusion of the experimental drug was started until the end of the operation, and the PCIA pump with the study medication is used during 2 days postoperatively.Continuous follow-up for three days after surgery.Follow-up personnel recorded LATCH score, VAS score, quality-of-recovery score and other indicators.In the 6th week after caesarean section, the outcome indicators were collected by electronic questionnaire and telephone follow-up.This randomized controlled trial is aims to prove that dexmedetomidine, used in parturient with elective cesarean section, can improve maternal mood and prolong the duration of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I or II
2. BMI≦35kg/m2
3. Greater than 37 weeks gestation
4. Expressed a desire to breastfeed for a least 3 months postpartum
5. Elective cesarean section

Exclusion Criteria:

1. Intraspinal anesthesia contraindication
2. Twin or fetal Intrauterine distress
3. Preoperative history of application of analgesia or sedative drug
4. Severe cardiac and pulmonary dysfunction
5. History of neurological and psychiatric diseases

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Parturients are females.
Enrollment: 160 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Postpartum depression at sixth week after caesarean section | 6th week postpartum
  The Edinburgh Postnatal Depression Scale(EPDS) was used to determine the presence of postpartum depression through an electronic questionnaire in the sixth week after delivery.
  The Edinburgh Postnatal Depression Scale(EPDS) consists of 10 items. According to the severity of the symptoms, each item is scored in 4 levels (0, 1, 2, 3 points) with a cumulative maximum score of 30 points.In order to reduce the rate of missed diagnosis, we refer to the previous literature and use 10 points as the diagnostic threshold for postpartum depression. A score of 10 or more is considered as postpartum depression.
Self-reported exclusive breastfeeding at sixth week after caesarean section | 6th week postpartum
  Self-reported exclusive breastfeeding at sixth week postpartum by telephone follow-up.If exclusive breastfeeding is discontinued, obtain the point of discontinuation.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale(HADS) score | Preoperative, 1st day and 2nd day postpartum
  Referring to the preoperative HADS score, the HADS on the second day after caesarean section were analyzed to judge the maternal emotional changes.
  The Hospital Anxiety and Depression Scale (HADS) includes two subscales of anxiety and depression, 7 questions per subscale, and 14 questions in total.Each question is divided into 4 score levels according to the severity (0, 1, 2, 3 points). The anxiety and depression subscales all use 8 points as the diagnostic threshold, and 8 or more points are considered to have anxiety or depression.
  The statistical analysis of this outcome indicator is mainly to regard the scale score as a continuous variable rather than a binary variable.
LATCH breastfeeding assessments | 1st day postpartum
  Day-1 LATCH (Latch, Audible swallowing, Type of nipple, Comfort, and Hold/help) breastfeeding assessments.
VAS score after cesarean section | 6,12,24 and 48 hours after cesarean section
  The basic method of Visual Analogue Scale(VAS) is to use a ruler with a length of about 10 cm, the ruler is marked with 10 scales, and the ends are "0" and "10" respectively. "0" indicate no pain, and "10" indicate unbearable pain. Ask the parturient to mark the position on the ruler that represents her pain level. Follow-up personnel record pain scores based on the location of the marker.
Quality-of-recovery score | Preoperative, 1st day and 2nd day postpartum
  Recovery quality assessment on the second day after delivery via the ObsQoR-11 scale.
  The ObsQoR-11 scale focuses on the following 11 items: nausea or vomiting, shivering, dizzy, in control, comfortable, able to hold baby, mobilising alone, personal hygiene, able to feed/nurse baby, moderate pain and severe pain. According to different degrees, each item can be divided into 0-10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Yan, M.D/Ph.D, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Result] Xu H, Ding Y, Ma Y, Xin X, Zhang D. Cesarean section and risk of postpartum depression: A meta-analysis. J Psychosom Res. 2017 Jun;97:118-126. doi: 10.1016/j.jpsychores.2017.04.016. Epub 2017 Apr 24. PMID 28606491
- [Result] Silva CS, Lima MC, Sequeira-de-Andrade LAS, Oliveira JS, Monteiro JS, Lima NMS, Santos RMAB, Lira PIC. Association between postpartum depression and the practice of exclusive breastfeeding in the first three months of life. J Pediatr (Rio J). 2017 Jul-Aug;93(4):356-364. doi: 10.1016/j.jped.2016.08.005. Epub 2016 Dec 26. PMID 28034730
- [Result] Hobbs AJ, Mannion CA, McDonald SW, Brockway M, Tough SC. The impact of caesarean section on breastfeeding initiation, duration and difficulties in the first four months postpartum. BMC Pregnancy Childbirth. 2016 Apr 26;16:90. doi: 10.1186/s12884-016-0876-1. PMID 27118118
- [Result] Nie Y, Liu Y, Luo Q, Huang S. Effect of dexmedetomidine combined with sufentanil for post-caesarean section intravenous analgesia: a randomised, placebo-controlled study. Eur J Anaesthesiol. 2014 Apr;31(4):197-203. doi: 10.1097/EJA.0000000000000011. PMID 24463478
- [Result] Yoshimura M, Kunisawa T, Suno M, Sugawara A, Kurosawa A, Nakanishi R, Aoki K, Toriumi T. Intravenous dexmedetomidine for cesarean delivery and its concentration in colostrum. Int J Obstet Anesth. 2017 Nov;32:28-32. doi: 10.1016/j.ijoa.2017.05.002. Epub 2017 May 10. PMID 28687146
- [Result] Schnabel A, Meyer-Friessem CH, Reichl SU, Zahn PK, Pogatzki-Zahn EM. Is intraoperative dexmedetomidine a new option for postoperative pain treatment? A meta-analysis of randomized controlled trials. Pain. 2013 Jul;154(7):1140-9. doi: 10.1016/j.pain.2013.03.029. Epub 2013 Mar 27. PMID 23706726
- [Result] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408
- [Result] Funai Y, Pickering AE, Uta D, Nishikawa K, Mori T, Asada A, Imoto K, Furue H. Systemic dexmedetomidine augments inhibitory synaptic transmission in the superficial dorsal horn through activation of descending noradrenergic control: an in vivo patch-clamp analysis of analgesic mechanisms. Pain. 2014 Mar;155(3):617-628. doi: 10.1016/j.pain.2013.12.018. Epub 2013 Dec 16. PMID 24355412
- [Result] Lau Y, Wang Y, Yin L, Chan KS, Guo X. Validation of the Mainland Chinese version of the Edinburgh Postnatal Depression Scale in Chengdu mothers. Int J Nurs Stud. 2010 Sep;47(9):1139-51. doi: 10.1016/j.ijnurstu.2010.02.005. Epub 2010 Mar 12. PMID 20219196
- [Derived] Wang Y, Fang X, Liu C, Ma X, Song Y, Yan M. Impact of Intraoperative Infusion and Postoperative PCIA of Dexmedetomidine on Early Breastfeeding After Elective Cesarean Section: A Randomized Double-Blind Controlled Trial. Drug Des Devel Ther. 2020 Mar 11;14:1083-1093. doi: 10.2147/DDDT.S241153. eCollection 2020. PMID 32210537